CLINICAL TRIAL: NCT05391893
Title: Emergency Department Atrial Fibrillation Oral Diltiazem Observation Protocol
Brief Title: Effect of Oral and Intravenous Diltiazem Protocol for Emergency Department Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGME#03-2021
Record Dates: First submitted 2021-09-23; First posted 2022-05-26 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Infusion Pumps

STUDY DESIGN:
Intervention Model Description: A treatment protocol using oral and IV diltiazem has been implemented. We will compare admission rates, time to heart rate control, and hypotension between the protocol group and patients receiving traditional treatments for atrial fibrillation with rapid ventricular response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diltiazem with oral and intravenous treatment (Active Comparator): Diltiazem 0.25mg/kg injection, give over 2 minutes, max dose 30mg. 15 minutes following Diltiazem Infusion administer oral Diltiazem 60mg IR Tablet, do not give if BP<100
  Interventions: Drug: Oral
- traditional atrial fibrillation with rapid ventricular response (Placebo Comparator): these patients will receive traditional treatments at provider discretion. To be included in teh study their initial heart rate must also be over 125, and they must receive at least one intravenous medication for atrial fibrillation with rapid ventricular response. This will be a heterogenous group of patients receiving digoxin, amiodarone, various beta-blockers, and intravenous diltiazem without oral diltiazem.
  Interventions: Drug: Intravenous drug

INTERVENTIONS:
Drug: Oral — Diltiazem 0.25mg/kg injection, give over 2 minutes, max dose 30mg
  Other Names: these patients will receive oral and intravenous diltiazem
  Arms: Diltiazem with oral and intravenous treatment
Drug: Intravenous drug — these patients will receive traditional treatments at provider discretion. They must receive at least one intravenous medication for atrial fibrillation with rapid ventricular response. This will be a heterogenous group of patients receiving digoxin, amiodarone, various beta-blockers, and intravenous diltiazem without oral diltiazem.
  Arms: traditional atrial fibrillation with rapid ventricular response

SUMMARY:
The primary objective of the study is to reduce hospital admission and decrease time to disposition through establishing an effective treatment protocol for AF and Atrial Flutter in the Emergency Department of Spectrum Health Lakeland. Secondary outcome is to measure if oral diltiazem is an effective HR controlling agent in AF RVR and Flutter.

ELIGIBILITY:
Inclusion Criteria:

* Heart rate >125
* Systolic BP>110
* Atrial Fibrillation/Flutter confirmed on ECG.
* Meets observation unit requirements (performs certain ADL's (acts of daily living)
* Age>18.

Exclusion Criteria:

* Wolf-Parkinson-White syndrome
* ST Elevation Myocardial Infarction
* Pregnant
* Clinical diagnosis of Sepsis,
* Decompensated HF
* allergy to Diltiazem
* provider discretion
* clinical need for cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Matthew Hysell, Saint Joseph, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diltiazem With Oral and Intravenous Treatment | Traditional Atrial Fibrillation With Rapid Ventricular Response
Started | 177 | 267
Completed | 172 | 249
Not Completed | 5 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diltiazem With Oral and Intravenous Treatment | Traditional Atrial Fibrillation With Rapid Ventricular Response | Total
Number analyzed (Participants) | 177 | 267 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (13.3) | 71 (12.7) | 70.05 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 138 | 240
  Male | 75 | 129 | 204
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 37 | 57
  White | 157 | 230 | 387
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 177 | 267 | 444

OUTCOME MEASURES:

1. Primary Outcome: Admission Rate
Description: This will compare rates of patients admitted between the protocol group and patients treated traditionally
Time Frame: 1 days
Measure: Count of Participants; unit: Participants
Arm/Group | Diltiazem With Oral and Intravenous Treatment | Traditional Atrial Fibrillation With Rapid Ventricular Response
Number analyzed (Participants) | 172 | 249
Participants | 98 | 188

2. Primary Outcome: Treatment Success at 3 Hours
Description: This will compare the total number of patients who in 3 hours from first medicine administration achieved heart rate less than 110 between the protocol and traditional treatment group
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Diltiazem With Oral and Intravenous Treatment | Traditional Atrial Fibrillation With Rapid Ventricular Response
Number analyzed (Participants) | 177 | 267
Participants | 150 | 192

3. Secondary Outcome: Rate of Hypotension
Description: rates of patients experiencing systolic blood pressure less than 90
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Diltiazem With Oral and Intravenous Treatment | Traditional Atrial Fibrillation With Rapid Ventricular Response
Number analyzed (Participants) | 177 | 267
Participants | 7 | 17

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 24 hours following emergency room admittance.
Arm/Group | Diltiazem With Oral and Intravenous Treatment | Traditional Atrial Fibrillation With Rapid Ventricular Response
All-Cause Mortality (participants affected / at risk) | 0/177 | 1/267
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/267
Other Adverse Events (participants affected / at risk) | 7/177 | 17/267
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diltiazem With Oral and Intravenous Treatment (N=177) | Traditional Atrial Fibrillation With Rapid Ventricular Response (N=267)
Hypotension (Vascular disorders) | 7 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT05391893/Prot_SAP_000.pdf